CLINICAL TRIAL: NCT00002742
Title: A PROSPECTIVE RANDOMIZED, DOUBLE-BLIND, COMPARATIVE, MULTICENTER STUDY TO EVALUATE EFFICACY AND SAFETY OF NYSTATIN AND AMPHOTERICIN B FOR EMPIRIC ANTIFUNGAL TREATMENT IN NEUTROPENIC PATIENTS
Brief Title: Antifungal Therapy for Fever and Neutropenia in Patients Receiving Treatment for Hematologic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aronex Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000064660; AR-95-41.356-006; NCI-V96-0845
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Myeloproliferative Disorders; Infection; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult Hodgkin lymphoma; adult non-Hodgkin lymphoma; leukemia; childhood non-Hodgkin lymphoma; chronic myeloproliferative disorders; myelodysplastic syndromes; childhood Hodgkin lymphoma; recurrent adult non-Hodgkin lymphoma; infection; multiple myeloma and other plasma cell neoplasms; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Infections; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — amphotericin B, deoxycholate drug combination; Nystatin

INTERVENTIONS:
Drug: amphotericin B deoxycholate
Drug: nystatin

SUMMARY:
RATIONALE: Antifungal therapy with liposomal nystatin may reduce fever and neutropenia in patients undergoing treatment for hematologic cancer. It is not yet known whether liposomal nystatin is more effective than standard amphotericin B in treating patients with fever and neutropenia who are receiving chemotherapy for hematologic cancer or bone marrow transplantation for leukemia.

PURPOSE: Randomized phase III trial to study the effectiveness of liposomal nystatin compared with standard amphotericin B to treat fever and neutropenia in patients receiving chemotherapy for hematologic cancer or bone marrow transplantation for leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of liposomal nystatin vs standard amphotericin B for the empiric treatment of persistent febrile neutropenic patients. II. Compare the incidence of drug-related toxicity or impairment and infusion-related toxicity in patients treated with liposomal nystatin vs standard amphotericin B. III. Determine the pharmacokinetics of liposomal nystatin.

OUTLINE: Randomized, double-blind study. Arm I: Antifungal Therapy. Liposomal Nystatin. Arm II: Antifungal Therapy. Amphotericin B, NSC-527017.

PROJECTED ACCRUAL: 350 evaluable patients will be studied in this multicenter trial.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Persistent febrile neutropenia associated with 1 of the following within 3 months prior to entry: Cytotoxic chemotherapy Bone marrow transplantation Neutropenia defined as either: ANC no greater than 500/mm3 ANC no greater than 1,000/mm3 and expected to decrease to 500/mm3 or less within 2 days after entry Persistent continuous or spiking fever of at least 38 C No association with administration of pyrogenic substances No response to at least 72 hours of empiric, broad-spectrum antibacterial therapy No microbiologically documented source of infection At least 30 days since documented invasive fungal infection

PATIENT CHARACTERISTICS: Age: 2 and over Performance status: Not specified Life expectancy: At least 28 days Hematopoietic: Not specified Hepatic: No grade 2 or greater hepatic impairment Renal: No grade 2 or greater renal impairment No peritoneal dialysis or hemodialysis Other: No history of severe allergic reaction to polyene antifungal agent No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile women during and for 3 months after study

PRIOR CONCURRENT THERAPY: At least 2 weeks since polyene antifungal therapy Concurrent oral prophylactic antifungal therapy with an azole antifungal agent (e.g., fluconazole, itraconazole) allowed if patient remains febrile No concurrent azole therapy At least 30 days since other investigational drug or device except investigational formulation of amphotericin B

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-01; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Gordon, MD, Study Chair — Aronex Pharmaceuticals
Locations (59):
- United States (59):
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Holt-Krock Clinic, Fort Smith, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Office of Rosalda Rodriguez, M.D., Chula Vista, California
  - Beckman Research Institute, City of Hope, Duarte, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - University of Colorado Cancer Center, Denver, Colorado
  - New Britain General Hospital, New Britain, Connecticut
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Tampa Children's Hospital, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - St. John's Pavilion - Springfield Clinic Research Department, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lake Charles Medical and Surgical Clinic, Lake Charles, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - United Hospital, Saint Paul, Minnesota
  - Columbia Comprehensive Cancer Care Clinic, Columbia, Missouri
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Antibiotic Research Associates, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore Cancer Center, Neptune City, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - St. Vincent's Medical Center of Richmond, Staten Island, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Brookview Research, Inc., Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Office of Ian Baird & Mark Herbert, Columbus, Ohio
  - Infectious Disease Associates of N.W. Ohio, Toledo, Ohio
  - Northeast Ohio Infectious Disease Associates, Inc., Youngstown, Ohio
  - Medical Specialists, Inc., Zanesville, Ohio
  - University of Oklahoma - Department of Pharmacy Practice, Oklahoma City, Oklahoma
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center at Knoxville, Knoxville, Tennessee
  - Baptist Clinical Research Services, Memphis, Tennessee
  - Texas Cancer Center at Brackenridge Hospital, Austin, Texas
  - University of Texas Southwestern Medical School, Dallas, Texas
  - Infectious Disease Associates of Houston, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Scott and White Clinic, Temple, Texas
  - Infections Limited, P.S., Tacoma, Washington